CLINICAL TRIAL: NCT00318799
Title: A Single-centre, Open-label, Crossover, Controlled, Randomized Study to Investigate the Impact of SH T00658ID as Compared to a Monophasic Contraceptive Containing Ethinylestradiol and Levonorgestrel (SH D01155E) on Hemostatic Parameters in 30 Healthy Female Volunteers Over 3 Treatment Cycles
Brief Title: Impact of SH T00658ID as Compared to a Monophasic Contraceptive Containing Ethinylestradiol and Levonorgestrel (SH D01155E) on Hemostatic Parameters
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 91477; 2005-004688-45 (EudraCT Number); 310122 (Other: Company internal)
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Pregnancy, Unplanned
Keywords: prevention of unintended pregnancies

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: EV/DNG (Qlaira, BAY86-5027, SH T00658ID)
- Arm 2 (Active Comparator)
  Interventions: Drug: SH D01155E

INTERVENTIONS:
Drug: EV/DNG (Qlaira, BAY86-5027, SH T00658ID) — per cycle (28 days): Days 1-2: 3.0 mg EV; Days 3-7: 2.0 mg EV + 2.0 mg DNG; Days 824: 2.0 mg EV + 3.0 mg DNG; Days 25-26: 1.0 mg EV; Days 27-28: Placebo
  Arms: Arm 1
Drug: SH D01155E — per cycle: Days 1-21: 0.03 mg EE + 0.15 mg LNG; Days 22-28: Placebo
  Arms: Arm 2

SUMMARY:
The aim of this study is to evaluate the impact of SH T00658ID (EV/DNG tablet) on hemostatic parameters in comparison to a reference oral contraceptive (OC) (SH D01155E) in a crossover design.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers

Exclusion Criteria:

* Pregnancy or lactation
* Any condition that might interfere with the outcome as all contraindications for OC use.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Intraindividual absolute changes from Baseline in the Parameters of thrombin and fibrin turnover | Baseline, Cycle 3 of each treatment period

SECONDARY OUTCOMES:
Intraindividual absolute changes from Baseline in Pro- and anti-coagulatory parameters and the parameter of thrombin and fibrin turnover (activation marker): Prothrombin (Factor II). | Baseline, Cycle 3 of each treatment period
Adverse events | 2 treatment periods (3 cycles each), 2 cycles whash out-period and 14 days follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Dinox B.V., Groningen, Netherlands

REFERENCES:
- [Result] Klipping C, Duijkers I, Parke S, Mellinger U, Serrani M, Junge W. Hemostatic effects of a novel estradiol-based oral contraceptive: an open-label, randomized, crossover study of estradiol valerate/dienogest versus ethinylestradiol/levonorgestrel. Drugs R D. 2011;11(2):159-70. doi: 10.2165/11591200-000000000-00000. PMID 21679006